CLINICAL TRIAL: NCT01960361
Title: A Multi-center Study to Evaluate Bone Loss, Survival Rate and Stability of ICE Implant System Over 24 Months, for Patients With Tooth Loss Requiring up to 4 Implants, in Staged Loading Protocol
Brief Title: A Multi-center Study to Evaluate Bone Loss, Survival Rate and Stability of ICE Implant
Acronym: ICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alpha - Bio Tec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICE_001
Record Dates: First submitted 2013-10-09; First posted 2013-10-10 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Implant Clinical Survival; Dental Implant Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICE dental implant (Experimental): Subjects implanted with ICE implant
  Interventions: Device: ICE dental implant

INTERVENTIONS:
Device: ICE dental implant — ICE- Implant Classical Esthetic implant

SUMMARY:
The current prospective clinical study's aim is to determine ABT's ICE implant survival rate, crestal interproximal bone resorption during 24 months post implant insertion and to assimilate the drilling sequence during the clinical use of ICE implants.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over the age of 18 years who need implantation of 1-4 implants.
2. Patients who are able to understand the requirements of the study, and are willing and able to comply with its instructions and schedules.
3. Patients who had provided written informed consent to participate in the study prior to any study procedure.
4. Patients in general good health in the opinion of the principal investigator as determined by medical history and oral examination.

Exclusion Criteria:

1. Immediate loaded implants.
2. Treatment with anticoagulant drugs (INR under 1.8) or bisphosphonates.
3. Treatment with anticonvulsants drugs.
4. Untreated Periodontal disease and inability of the patient to maintain reasonable oral hygiene according to study requirements.
5. Patients with history of alcohol, narcotics or drug abuse.
6. Patients under steroid therapy.
7. Patients receiving radiotherapy, chemotherapy or any other immunosuppressive treatment or who have been administered radiotherapy in the last 5 years.

   Patients through at anytime received radiotherapy to the head and neck region will be excluded anyway.
8. Metabolic bone disorders and/or bone augmentation.
9. Uncontrolled bleeding disorders such as: hemophilia, thrombocytopenia, granulocytopenia.
10. Degenerative diseases.
11. Osteoradionecrosis.
12. Renal failure.
13. Organ transplant recipients.
14. HIV positive.
15. Malignant diseases.
16. Diseases that compromise the immune system.
17. Unbalanced diabetes mellitus. (HbA1c above 6.5)
18. Psychotic diseases.
19. Hypersensitivity to one of the components of the implant in general and titanium in particular.
20. Women who are pregnant or lactating.
21. Lack of patient cooperation.
22. Uncontrolled endocrine diseases.
23. Any systemic condition that is unbalanced and therefore precludes surgical procedures.
24. Parafunctional habits.- e.g Bruxism.
25. Temporomandibular joint disease.
26. Various pathologies of the oral mucosa for example: Benign mucous pemphigoid, desquamative ginigivitis, erosive lichen planus ,malignancy of oral cavity, bolus erosive diseases of the oral mucosa.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-03 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Cumulative Survival Rate | 24 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Rishon LeZiyyon, Israel